CLINICAL TRIAL: NCT01617733
Title: An Open Label, Longitudinal Study of the Effects of Subcutaneous Acute and Chronic Pasireotide (som230) Therapy on Adrenocorticotrophic Hormone and Tumour Volume in Patients With Nelson's Syndrome
Brief Title: Pasireotide Therapy in Patients With Nelson's Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate patient recruitment
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Novartis (Industry); The Christie NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH15164; 2009-014457-33 (EudraCT Number)
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Nelson Syndrome
MeSH Terms: conditions — Nelson Syndrome | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pasireotide (Experimental): 4 Weeks pasireotide 0.6mg s/c injections twice daily followed by 24 weeks treatment with pasireotide LAR 60mg every 28 days with dose reductions if poor tolerability is encountered
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Pasireotide — 4 Weeks pasireotide 0.6mg s/c injections twice daily followed by 24 weeks treatment with pasireotide LAR 60mg every 28 days with dose reductions if poor tolerability is encountered

SUMMARY:
Nelson's syndrome, an expanding pituitary tumour, occurs in up to 30% of adults after bilateral adrenalectomy for Cushing's disease, for which no medical treatment exists. Plasma Adrenocorticotrophic hormone (ACTH) levels in these patients remain high, they are characteristically deeply pigmented, and may experience neurological effects as a consequence of the tumour. It is not known whether the tumour growth is due to the lack of cortisol feedback after adrenalectomy or whether the pituitary cells were preprogrammed to develop into a tumour.

There is a real need for an effective medical management for Nelson's syndrome. This is especially true given the increasing data on the somewhat disappointing longterm outcome of transsphenoidal surgery, and the increasing use of aparoscopic bilateral adrenalectomy for failures of pituitary surgery or even as primary therapy for Cushing's disease. Therefore, it is likely that there will be increasing numbers of patients attending endocrine centres worldwide with Nelson's syndrome following bilateral adrenalectomy as part of their management for Cushing's disease. In view of this it is important to investigate all potential avenues for the treatment of Nelson's syndrome and translate any benefits to patients.

This study, designed and initiated by the investigators, will assess if pasireotide reduces ACTH levels and tumour volume in patients with Nelson's syndrome. Patients will be recruited for a period of 32 weeks and receive 4 weeks of pasireotide twice daily and then 24 weeks of pasireotide long acting release therapy every 4 weeks. Over the 32 week protocol patients will make 12 visits for serial ACTH blood measurements and have 2 MRI scans to assess tumour volume.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* To be verified at Visit one and confirmed at Visit two
* Male or female patients aged 18-80 years
* Signs and symptoms consistent with Nelson's Syndrome
* Biochemistry consistent with Nelsons syndrome: failure to suppress plasma ACTH to less than 200 pg/ml at 2 hours following morning dose of hydrocortisone
* Negative pregnancy test where applicable

Exclusion Criteria:

* Received any prior or current treatment with a pasireotide or other somatostatin analogue.
* Requires surgery for recent significant deterioration in visual fields or other neurological signs related to tumour mass.
* Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis, or persistent ALT, AST, alkaline phosphates 2X> upper limit of normal, or total bilirubin 1.5X> upper limit of normal.
* Patients with symptomatic cholelithiasis
* Abnormal clinical laboratory values considered by the Investigator to be clinically significant and which could affect the interpretation of the study results
* QTcF interval as measured by ECG >480msecs
* Any current or prior medical condition that may, in the opinion of the Investigator, interfere with the conduct of the study or evaluation of the results.
* Female patients who are pregnant or lactating, or of childbearing potential and not practising a medically acceptable method of birth control. Medically acceptable methods include including the oral contraceptive pill, intrauterine devices, mechanical methods (e.g. vaginal diaphragm, vaginal sponge, or condom with permicidal jelly).
* History of alcohol or drug abuse in the sixmonth period prior to Visit 1, or who plan to take an investigational
* History of alcohol or drug abuse in the six month period prior to Visit 1, or who plan to take an investigational drug for another study during this study.
* History of noncompliance to medical regimes or who are considered potentially unreliable.
* Pituitary radiotherapy within the last 1 year prior to study entry.
* Unable to complete the entire study for any reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-03; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Serum ACTH levels in patients with Nelson's syndrome. | 0, 2, 4, 8, 12, 16, 20, 24, 28 weeks
  Early morning plasma ACTH sampled at 0, 1, 2, and 3 hours after morning hydrocortisone (HC) during 4 weeks of pasireotide 1200ug/day compared with levels at these respective time points found at baseline, and after chronic depot pasireotide 60mg i.m every 28 days:
  Complete success: Fall in pre-HC plasma ACTH > 400ng/l, or 120 minutes after HC >200ng/l Partial success: Fall in pre-HC plasma ACTH < 399ng/l >200ng/l, or 120 minutes after HC <199ng/l >100ng/l No success: Fall in pre-HC plasma ACTH < 199ng/l, or 120 minutes after HC <99ng/l

SECONDARY OUTCOMES:
Tumour volume in patients with Nelson's syndrome. | 0 & 28 weeks
  Does Chronic Pasireotide Therapy Effect Tumour Volume?
  H0= Pasireotide will not reduce tumour volume in patients with Nelson's syndrome.
  H1= Pasireotide will reduce tumour volume in patients with Nelson's syndrome.
Is the Pasireotide Therapy Used in this Study Safe and Tolerable in Nelson's Patients? | 0, 2, 4, 8, 12, 16, 20, 24, 28 weeks
  Overall outcome measure
Does tumour volume correlate with somatostatin receptor expression? | 0 & 28 weeks
  Tumour volume from MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: John Newell-Price, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Barts and the London NHS Trust, London
  - The Christie Hospital NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Trust, Oxford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

REFERENCES:
- [Derived] Daniel E, Debono M, Caunt S, Girio-Fragkoulakis C, Walters SJ, Akker SA, Grossman AB, Trainer PJ, Newell-Price J. A prospective longitudinal study of Pasireotide in Nelson's syndrome. Pituitary. 2018 Jun;21(3):247-255. doi: 10.1007/s11102-017-0853-3. PMID 29313180